CLINICAL TRIAL: NCT06890897
Title: Effect of Intravenous Infusion of Esketamine Combined Pulsed Radiofrequency on Acute/Subacute Zoster-associated Trigeminal Neuralgia
Brief Title: Esketamine Combined Pulsed Radiofrequency for Acute/Subacute Zoster-associated Trigeminal Neuralgia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Beijing Xiaotangshan Hospital (Other); The First Hospital of Fangshan District,Beijing (Other); Beijing Ditan Hospital (Other); Hengshui People's Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Director of Department of Day surgery and Pain Management Affiliation, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY-2024-332-02-01
Record Dates: First submitted 2025-03-12; First posted 2025-03-24 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Zoster; Herpes, Trigeminal Neuralgia (Etiology)
Keywords: acute/subacute zoster-associated trigeminal neuralgia; esketamine; pulsed radiofrequency
MeSH Terms: conditions — Herpes Zoster; Herpes Simplex; Trigeminal Neuralgia | interventions — Esketamine; Prolactin-Releasing Hormone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esketamine group (Experimental): Besides PRF plus standardized treatment, patients will also receive intravenous infusion of Esketamine ;
  Interventions: Drug: Esketamine group
- control group (Active Comparator): Patients will only receive PRF plus standardized treatment
  Interventions: Drug: PRF group

INTERVENTIONS:
Drug: Esketamine group — Patients in the esketamine group will receive intravenous infusion of esketamine besides PRF+standardized treatment.The formula will be intravenous infusion of 0.5mg/kg of esketamine diluted in 50 mL normal saline, starting with intravenous injection of 10 mg of esketamine for 1 minute, and maintaining a dose 8 mg/h.The infusion rate will be adjusted the parameter according to the tolerance of the patients
  Other Names: Esketamine + PRF+standardized treatment
  Arms: Esketamine group
Drug: PRF group — Patients in the control group will receive PRF+standardized treatment
  Other Names: PRF + standardized group
  Arms: control group

SUMMARY:
To assess the 1-month effects and safety of esketamine combined PRF and standardized treatment to relieve pain in patients with acute/subacute zoster-related trigeminal neuralgia(ZRTN).

DETAILED DESCRIPTION:
The investigators aim to investigate whether or not esketamine combined PRF and standardized treatment to relieve pain in patients with acute/subacute ZRTN , and seek a safe, and effective treatment for refractory patients with ZRTN

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years;
2. History of HZ within the last three months;
3. Lesions located in the trigeminal nerve or its branches innervated regions；
4. Numeric Rating Scale (NRS) pain score≥4 (NRS, 0 = no pain, 10= worst possible pain) with pharmacotherapy;
5. Planned to perform CT-guided PRF treatment of the Gasserian ganglion .

Exclusion Criteria:

1. Obstructive sleep apnoea syndrome;
2. Those who receive other invasive treatments, such as spinal cord stimulation;
3. A history of systemic immune diseases, organ transplantation, or cancers;
4. A history of severe cardiopulmonary, hepatic or renal dysfunction;
5. A history of schizophrenia, epilepsy, or myasthenia gravis, delirium;
6. Comorbid hyperthyroidism or phaeochromocytoma;
7. Recent history of drug abuse;
8. Having contraindications to esketamine;
9. Communication difficulties.

Withdrawal criteria

1. Lost to follow-up during the study;
2. Not perform the planned operation;
3. Receiving other treatment regimes during the study period;
4. Not suitable for continuing the study for emerging severe comorbidities or special physiological changes during the study;
5. Voluntary withdrawal from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
the NRS score at 1 month after treatment. | 1-month period
  The Numeric Rating Scale (NRS) score is a way to quantify the degree of subjective feelings such as pain using numbers. Generally, 0 represents no pain, and 10 represents the most severe pain.A higher score indicates more severe pain

SECONDARY OUTCOMES:
the 12-item Short-Form Health Survey (SF-12) score | at 1 day, 1 week, 2 weeks, 1 month, 2 months, 3 months after treatment
  Quality of life (QoL) assessed by the SF-12 score (range 0-100, with higher scores indicating better health status)
the Pittsburgh Sleep Quality Index (PSQI) score | at 1 day, 1 week, 2 weeks, 1 month, 2 months, 3 months after treatment
  Sleep quality measured by PSQI score（range 0-21, with higher scores indicating poorer sleep quality）
the Patient Global Impression of Change scale (PGIC) | at 1 day, 1 week, 2 weeks, 1 month, 2 months, 3 months after treatment
  The proportion of patients with a response of "no change", "minimally improved", "much improved" or "very much improved" on PGIC
Analgesics consumption | at 1 day, 1 week, 2 weeks, 1 month, 2 months, 3 months after treatment
  the type of analgesics and analgesics consumption
Safety assessments | at 0 day, 1 day, 1 week, 2 weeks,1 month, 2 months, 3 months
  intraoperative complications, PRF-related complications, Eskatamine-related complications

CONTACTS AND LOCATIONS:
Overall Officials: Fang Luo, M.D., Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
Not yet